CLINICAL TRIAL: NCT03491358
Title: Inhaled Allergen Challenge Methodology: Assessment of a Vibrating Mesh Nebulizer for Allergen Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, College of Medicine, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SOLO ALLERGEN 18
Record Dates: First submitted 2018-03-29; First posted 2018-04-09 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Asthma
Keywords: vibrating mesh nebulizer; allergen challenge
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wright jet nebulizer (Active Comparator): Will employ the Wright jet nebulizer for use in an allergen challenge triad
  Interventions: Device: Wright jet nebulizer
- Solo vibrating mesh nebulizer (Experimental): Will employ the Aerogen Solo vibrating mesh device for use in an allergen challenge triad
  Interventions: Device: Aerogen Solo

INTERVENTIONS:
Device: Wright jet nebulizer — Roxon Medi-Tech, Montreal, QC, Canada
  Arms: Wright jet nebulizer
Device: Aerogen Solo — Aerogen Ltd., Galway, Ireland
  Arms: Solo vibrating mesh nebulizer

SUMMARY:
This study will assess the Aerogen Solo® (Solo®) vibrating mesh nebulizer as a potential new device for use in allergen challenge testing.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, cross-over study utilizing the expertise of three Canadian academic centers (University of Saskatchewan, McMaster University, Laval University) that have been performing allergen inhalation challenges and other bronchoprovocation studies for more than forty years.

Each participant will be required to attend the research lab on five occasions (Visits 1-5). At Visit 1, study staff will provide an overview of the study purpose and procedure and answer any questions the participant may have. The individual will then provide consent if they wish to participate (i.e. sign the consent form). Skin prick testing to determine relevant allergen sensitivities and to determine which allergen extract will be used for the skin test endpoint (STE) and allergen inhalation challenge will then be performed. The participant will be randomized with respect to which nebulizer (Solo® or Wright) will be used first. The choice of nebulizer for the first participant will be via blinded draw. Subsequent nebulizer assignments will alternate. Participants will undergo the STE procedure and methacholine challenge testing (MCT) at visit 2; an allergen challenge will be done the next day at Visit 3 using the same nebulizer as was used for the MCT at Visit 2. Visits 4 and 5 will also be performed on consecutive days and will involve methacholine and allergen challenge testing, respectively, using the nebulizer that was not used at Visits 2 and 3. A minimum of two weeks must separate Visits 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

* baseline FEV1 greater than or equal to 70%
* positive response to inhaled methacholine (i.e. PD20 less than 400mcg)
* evidence of atopy (i.e. positive skin prick test to an allergen that can be used for the inhalation challenge
* absence of respiratory infection for at least 4 weeks
* absence of allergen exposure (or other trigger of upper or lower respiratory symptoms) for at least 4 weeks
* current nonsmoker (ex-smoker allowed; case by case basis; investigator discretion)
* require only infrequent short-acting beta2 agonist (i.e. salbutamol or terbutaline) to treat/control asthma (i.e. no inhaled corticosteroid or combination therapies, no intranasal corticosteroid; anti-histamines etc.)
* general good health with no other medical condition, medication use or lifestyle activities that would influence the outcome of the allergen challenge

Exclusion Criteria:

* pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Allergen Solo EAR PD20 (provocative dose causing a 20% fall in forced expiratory volume, FEV1) | Baseline
  Record the dose of allergen required to induce a 20% fall in forced expiratory volume using the Solo device

SECONDARY OUTCOMES:
Predicted allergen Solo EAR PD20 | Baseline (based on baseline methacholine challenge and skin test endpoint results)
  Will be predicted using the standard equation that employs the STE and MCT results

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Laval University, Québec, Quebec
  - Asthma Research Lab - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cockcroft DW, Davis BE, Blais CM, Boulet LP, Boulay ME, Villeneuve H, Gauvreau GM, O'Byrne PM, Howie KJ, Obminski CD. Use of a vibrating mesh nebulizer for allergen challenge. Allergy Asthma Clin Immunol. 2019 Nov 26;15:73. doi: 10.1186/s13223-019-0392-8. eCollection 2019. PMID 31788006